CLINICAL TRIAL: NCT01417923
Title: The Immune and Clinical Impacts of Vitamin D in Patients With Chronic Musculo-skeletal Pain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0042-11-MMC
Record Dates: First submitted 2011-08-01; First posted 2011-08-16 (Estimated); Last update posted 2012-11-06 (Estimated); Status verified 2012-11

CONDITIONS: Vitamin D Deficiency; Chronic Pain Syndrome; Inflammatory Response
Keywords: chronic musculo-skeletal pain; therapeutic&serology effects of vitamin D; CRP, IL-6, IL-8, TNF and prostaglandin E2; patients suffering from chronic musculo-skeletal pain
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- vitamin D (Experimental): We enrolled 80 patients of the age 18-80 years suffering from chronic musculo-skeletal pain (low back pain, fibromyalgia, chronic widespread pain) at least 6 months. The 40 patients will receive daily doses of 4000 units of vitamin D for 6 weeks
  Interventions: Drug: vitamin D

INTERVENTIONS:
Drug: vitamin D — P.O.4000 units Vit D per day for 6 weeks
  Other Names: VIT D "SOLGAR"

SUMMARY:
Vitamin D3 is produced in the skin following exposure to UVB light from the sun or artificial sources, and occurs naturally in a small range of foods.More recently, several reports underlined the impact of vitamin D on the prevalence and consequences of inadequate vitamin D intake and the research supporting its benefits for alleviating chronic musculoskeletal pain and fatigue syndromes in outpatients. Experts have recommended that vitamin D inadequacy should be addressed in all patients with bone or joint pain, myalgia, fibromyalgia, or chronic fatigue syndrome. It appears that soothing the daily musculoskeletal pain by supplementation of vitamin D may be a simple, well tolerated, and cost-effective modality.

Aim of study:

To study the potential therapeutic effects of vitamin D supplementation on patients with persistent musculo-skeletal pain. Clinicalparameters, visual analog score,short form McGill Pain Questionnaire,patient global perceived effect, quality of life assessed by SF-36 Questionnaire and laboratory parameters, the levels of 25 OH-Vitamin D, CRP, IL-6, IL-8, TNF and prostaglandin E will be assessed.

DETAILED DESCRIPTION:
The immune and clinical impacts of vitamin D in patients with chronic musculo-skeletal pain

Background Vitamin D is a group of fat-soluble secosteroids, the two major physiologically relevant forms are vitamin D2 (ergocalciferol) and vitamin D3 (cholecalciferol). Vitamin D without a subscript refers to either D2 or D3 or both. Vitamin D3 is produced in the skin following exposure to UVB light from the sun or artificial sources, and occurs naturally in a small range of foods. Vitamin D is carried in the bloodstream to the liver, where it is converted into the prohormone calcidiol. Circulating calcidiol may then be converted into calcitriol, the biologically active form of vitamin D, either in the kidneys or by monocyte-macrophages in the immune system. When synthesized by monocyte-macrophages, calcitriol acts locally as a cytokine, defending the body against microbial invaders (1).

When synthesized in the kidneys, calcitriol circulates as a hormone, regulating among other things, the concentration of calcium and phosphate in the bloodstream, promoting the healthy mineralization, growth and remodeling of bone, and also vital to the normal function of the different arms of the immune system (1;2).

Vitamin D receptor activation in the intestine, bone, kidney, and parathyroid gland cells leads to the maintenance of calcium and phosphorus levels in the blood (with the assistance of parathyroid hormone and calcitonin) and to the maintenance of bone content. Vitamin D increases expression of the tyrosine hydroxylase gene in adrenal medullary cells. Vitamin D is involved in the biosynthesis of neurotrophic factors, synthesis of nitric oxide synthase, and increased glutathione levels. Adequate vitamin D may also be associated with healthy hair follicle growth cycles (3). Vitamin D insufficiency can result in thin and brittle bones, whereas sufficiency prevents rickets in children and osteomalacia in adults and helps to protect elderly from osteoporosis. Vitamin D has also direct on muscle strength and function (4;5). Nevertheless, there is no persuasive evidence of lower vitamin D status in chronic pain sufferers.

There are also associations between low 25(OH)D levels and peripheral vascular disease (6), certain cancers (7-10), multiple sclerosis (11), rheumatoid arthritis (12-15), juvenile diabetes (16-18), Parkinson's and Alzheimer's disease (19;20). However these associations were found in observational studies and vitamin D vitamin supplements have not been demonstrated to reduce the risks of these diseases.

More recently, several reports underlined the impact of vitamin D on the prevalence and consequences of inadequate vitamin D intake and the research supporting its benefits for alleviating chronic musculoskeletal pain and fatigue syndromes in outpatients. There are extensive reports of pain worldwide and much of it is chronic, lasting 3 or more months, primarily involving muscles, bones and joints. In the United States, more than half of all adults participating in surveys have reported long term persistent or intermittent pain, with the lower and upper back, neck, shoulders, hips, and knees mentioned most frequently (21). For lower-back pain alone, an annual incidence of 50% and a lifetime prevalence of up to 80% have been reported (22). In more than 8 out of 10 cases, the causes are nonspecific, without evidence of injury, disease, or anatomical defect (23;24). More than a quarter (28%) of patients with chronic pain rate the effectiveness of medical treatments as poor, and most (77%) believe that new options are needed to treat their pain (25-27). It appears that soothing the daily musculoskeletal pain by supplementation of vitamin D may be a simple, well tolerated, and cost-effective modality. Experts have recommended that vitamin D inadequacy should be addressed in all patients with bone or joint pain, myalgia, fibromyalgia, or chronic fatigue syndrome (28;29). However, this seems to be unknown or overlooked by many healthcare providers. Research on vitamin D is still an emerging field, and there are divergent opinions among experts regarding many aspects of vitamin D pharmacology, function, and adequate intake needed for good health. While further research is needed, the clinical evidence to date recommending vitamin D supplementation for musculoskeletal pain and associated symptoms seems to be growing. In 3670 patients taking part in different studies with musculoskeletal pain significant vitamin D inadequacies were found in 48% to 100%. A study from the Mayo Clinic reported that a whopping 93% of patients with "chronic nonspecific pain syndromes" had deficient levels of vitamin D (30). When supplementation was provided for improving vitamin D status, pain and/or muscle weakness were resolved or at least subsided in most cases, and there were associated improvements in physical functioning.

A recently reported prospective study of 51 patients with type 2 diabetes and associated chronic, painful neuropathy found that conservative vitamin D supplementation (about 2000 IU/day) for 3 months resulted in nearly a 50% decrease in pain scores, with symptoms improving from "distressing" to "mild" on average (31). There had been an earlier case report of a patient with type 1 diabetes whose severe neuropathy had confined her to a wheelchair. This patient's aches and pains were resolved by high-dose vitamin D supplementation, and she reportedly was able to walk unassisted within 4 weeks (32). Other therapies need not be discontinued during a trial of vitamin D "analgesia.

Miller et al (33) evaluated in a cohort from the Baltimore Hip Studies, women aged >65 years were at baseline and 2, 6, and 12 months after hip fracture repair. Serum at baseline was analyzed for 25-hydroxyvitamin D [25(OH)D] and serum from all time points was analyzed for IL-6, women with vitamin D deficiency at the time of hip fracture had higher serum IL-6 levels in the year after hip fracture.

Aim of study To study the potential therapeutic effects of vitamin D supplementation on patients with persistent musculo-skeletal pain. Clinical and laboratory parameters will be assessed.

Methods We enrolled 80 patients of the age 18-80 years suffering from chronic musculo-skeletal pain (low back pain, fibromyalgia, chronic widespread pain) at least 6 months. The enrollees will be randomized in a double-blinded manner into the two following groups: Group 1 will receive daily doses of 4000 units of vitamin D ( 4 drops of 1,000 each) and Group 2 will receive a placebo. Written informed consent will be obtained from all participating patients.

On the day of recruitment blood will be drawn in order to determine the levels of 25 OH-Vitamin D, CRP, IL-6, IL-8, TNF and prostaglandin E2. Vitamin D or placebo will be taken for 6 weeks on top of the individual's daily medications. A second blood analysis will be conducted following the 6 week duration.

Additional outcome measures pain intensity assessed by visual analog score (VAS) (0 = no pain, 10 = worst imaginable pain), short form McGill Pain Questionnaire (SMPQ), patient global perceived effect (PGPE), scored by the patient on a 7-point Likert scale (from very bad to very good), quality of life assessed by SF-36 Questionnaire will be evaluated at base line, 6 weeks, 12 weeks and 6 months after the inclusion . At 12 weeks period a third 25 OH-Vitamin D blood level will be measured. Rescue medication will be provided as paracetamol 325mg+codein 15 mg. Consumption of pain medication will be recorded during the study and 2 week intervals. Adverse events will be recorded on each 6 weeks period and on patient report.

The vitamin D levels will be assessed by using the commercial kit, LIAISON® 25-OH vitamin D Assay (310900) (Cardinal Health, Inc., Dublin, OH, USA). The method for quantitative determination of 25-OH vitamin D is a direct, competitive chemiluminescence immunoassay.

The other assays will be assessed by ELISA kits. Statistics will be performed using the SPSS 18th edition using the Student's t-test or the Chi-Square test and if appropriate with Fisher's exact test. To adjust for differences in the baseline values, the analyses will be performed by using a multivariate logistic regression model. Consumption of medication will be compared using the Man-Whitney U test. Significance will be regarded if the p values will be lower than 0.05.

ELIGIBILITY:
Inclusion Criteria:

* We enrolled patients suffering from chronic musculo-skeletal pain (low back pain, fibromyalgia, chronic widespread pain) at least 6 months.

Exclusion Criteria:

* Patients with low compliance
* Allergy for vit D

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
serologic inflamatory responses with prolong vitamin D therapy | 6 weeks
  On the day of recruitment blood will be drawn in order to determine the levels of 25 OH-Vitamin D, CRP, IL-6, IL-8, TNF and prostaglandin E2. Vitamin D or placebo will be taken for 6 weeks on top of the individual's daily medications. A second blood analysis will be conducted following the 6 week duration

CONTACTS AND LOCATIONS:
Overall Officials: Meir Bennun, MD, Principal Investigator — Israel:Clalit Health Services, Meir Medical Center, PAIN CLINIC
Locations (1):
- Meir Medical Center, Kfar Saba, Israel